CLINICAL TRIAL: NCT05055089
Title: Short- and Medium-term Outcomes of New Generation Biological Aortic Valves in Aortic Valve Replacement Surgery
Brief Title: Short- and Medium-term Results of New Generation Aortic
Acronym: RVANG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0186
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Echocardiography; Aortic Valve; Cardiac Surgery; Mortality
Keywords: Echocardiography; Aortic valve; New-generation bioprosthesis; Conventional bioprosthesis; Rapid-deployment bioprosthesis; Sutureless valves; Function prostheses; Cardiac Surgery; Mortality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- new-generation bioprostheses: Patients undergoing surgical aortic valve replacement with new-generation bioprostheses
- traditional bioprosthesis: patients who received a traditional bioprosthesis

SUMMARY:
Over the past decade, aortic valve replacement surgery has undergone significant changes in terms of both the approaches and the prostheses used. In parallel with the historical biological prostheses for aortic valve surgery, a new generation of bioprostheses has been marketed since 2008, with the entry of these new prostheses in the armatorium of the Amiens-Picardy University Hospital since 2010. These are rapid deployment prostheses or prostheses without sutures. As a result, patients undergoing aortic valve replacement have been able to benefit from this type of bioprosthesis during their procedures. There are few publications reporting the 5-year follow-up of these bioprostheses. The investigators therefore decided to follow up patients operated on by a new generation bioprosthesis to study the 5-year survival and the functioning of their bioprostheses, in order to make a scientific contribution to the follow-up of these valves. These patients will be compared to patients who have benefited from the implantation of traditional bioprostheses.

ELIGIBILITY:
Inclusion Criteria:

* Retrospectively included all patients examined since 2010.
* Patients who have aortic valve surgery from the Cardiac Surgery Department of the University Hospital of Amiens.

Exclusion Criteria:

* Refusal to participate in the patient.
* Patients who have previously had aortic valve surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Cardiac Surgery Department of the University Hospital of Amiens of Picardy, France, short- and medium-term survival of patients undergoing surgical aortic valve replacement with new-generation bioprostheses compared with patients who received a traditional bioprosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Variation of mortality rate between both groups | 3 months
  both groups are :
  * Patients undergoing surgical aortic valve replacement with new-generation bioprostheses
  * Patients who received a traditional bioprosthesis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Nord, Amiens, France

IPD SHARING:
Plan to Share IPD: No